## STATISTICAL ANALYSIS PLAN FOR CLINICAL STUDY REPORT

A SINGLE-ARM, OPEN-LABEL PHASE 2 STUDY OF NIVOLUMAB (BMS-936558) IN SUBJECTS WITH RELAPSED OR REFRACTORY FOLLICULAR LYMPHOMA (FL) (CHECKMATE 140: CHECKPOINT PATHWAY AND NIVOLUMAB CLINICAL TRIAL EVALUATION 140)

PROTOCOL CA209-140

VERSION # 3.1

# **TABLE OF CONTENTS**

| STATIS | TICAL ANALYSIS PLAN FOR CLINICAL STUDY REPORT | 1 |
|---------|------------------------------------------------------|----|
| TABLE | OF CONTENTS | 2 |
| LIST OF | F TABLES | 5 |
| LIST OF | F FIGURES | 5 |
| 1 | BACKGROUND AND RATIONALE | 6 |
| 2 | STUDY DESCRIPTION | 8 |
| 2.1 | Study Design | 8 |
| 2.2 | Treatment Assignment | 9 |
| 2.3 | Blinding and Unblinding | 9 |
| 2.4 | Protocol Amendments | 9 |
| 2.5 | Data Monitoring and Other External Committees | 10 |
| 3 | OBJECTIVES | 10 |
| 3.1 | Primary objective | 10 |
| 3.2 | Secondary objectives | 10 |
| 3.3 | Exploratory Objectives | 11 |
| 4 | ENDPOINTS | 11 |
| 4.1 | Primary endpoint ORR (IRRC-assessed) | 11 |
| 4.2 | Secondary Endpoints | 12 |
| 4.2.1 | Duration of Response (IRRC-assessed) | 12 |
| 4.2.2 | Complete Remission Rate and Duration (IRRC-assessed) | 13 |
| 4.2.3 | Partial Remission Rate and Duration (IRRC-assessed) | 13 |
| 4.2.4 | Progression Free Survival (IRRC-assessed) | 13 |
| 4.2.5 | Objective Response Rate (Investigator-assessed) | 14 |
| 4.3 | Exploratory Endpoints | 15 |
| 4.3.1 | Safety and Tolerability | 15 |
| 4.3.1.1 | Immune-Mediated Adverse Events | 15 |
| 4.3.2 | Progression Free Survival (investigator-assessed) | 15 |
| 4.3.3 | Overall Survival | 15 |
| 4.3.4 | Other efficacy endpoints | 15 |
| 4.3.5 | Pharmacokinetics | 16 |
| 4.3.6 | Immunogenicity | 16 |
| 4.3.7 | Outcome Research | 16 |

| 4.3.7.1 | EORTC-QLQ-C30 | 16 |
|---|---|---|
| 4.3.7.2 | EuroQoL EQ-5D | 17 |
| 4.3.8 | Biomarker Data | 18 |
| 4.3.8.1 | PD-L1 Expression per Dako IHC assay | 18 |
| 4.3.8.2 | Other Biomarkers | 18 |
| 5 | SAMPLE SIZE AND POWER | 19 |
| 6 | STUDY PERIODS, TREATMENT REGIMENS AND POPULATIONS FOR ANALYSES | 19 |
| 6.1 | Study Periods | 19 |
| 6.1.1 | Baseline Period | 19 |
| 6.1.2 | Post Baseline Period | 20 |
| 6.2 | Treatment Regimens | 20 |
| 6.3 | Populations for Analyses | 20 |
| 6.3.1 | Analysis Populations | 20 |
| 7 | STATISTICAL ANALYSES | 21 |
| 7.1 | General Methods | 21 |
| 7.2 | Study Conduct | 21 |
| 7.2.1 | Accrual | 21 |
| 7.2.2 | Relevant Protocol Deviations | 21 |
| 7.3 | Study Population | 22 |
| 7.3.1 | Subject Disposition | 22 |
| 7.3.2 | Demographics and Other Baseline Characteristics | 22 |
| 7.3.3 | Medical History | 23 |
| 7.3.4 | Prior therapy | |
| 7.3.5 | Baseline Examinations | 23 |
| 7.4 | Extent of Exposure | 23 |
| 7.4.1 | Administration of Study Therapy | 23 |
| 7.4.2 | Modifications of Study Therapy | 24 |
| 7.4.2.1 | Dose delays | 24 |
| 7.4.2.2 | Infusion Interruptions and Rate Changes | 24 |
| 7.4.2.3 | Dose Reductions/Escalation | 25 |
| 7.4.3 | Concomitant Medications | 25 |
| 7.5 | Efficacy | 25 |

| 7.5.1 | Primary endpoint of ORR (IRRC-assessed) | 25 |
|---|---|---|
| 7.5.1.1 | ORR Subgroups | |
| 7.5.1.2 | Sensitivity analyses for ORR | 26 |
| 7.5.2 | Secondary Endpoint of Duration of Response (IRRC-assessed) | 26 |
| 7.5.3 | Secondary Enpoint of Complete Remission Rate (IRRC-assessed) | 26 |
| 7.5.4 | Secondary Endpoint of Partial Remission Rate and Duration (IRRC-assessed) | 27 |
| 7.5.5 | Secondary Endpoint of Progression Free Survival (IRRC-assessed) | |
| 7.5.6 | Secondary Endpoint of Objective Response Rate (Investigator-assessed) | 28 |
| 7.5.7 | Exploratory Endpoints | 28 |
| 7.5.7.1 | Progression Free Survival (investigator-assessed) | 28 |
| 7.5.7.2 | Overall Survival | 28 |
| 7.5.7.3 | Other efficacy analysis | 29 |
| 7.6 | Safety | 30 |
| 7.6.1 | Deaths | 30 |
| 7.6.2 | Serious Adverse Events | 30 |
| 7.6.3 | Adverse Events Leading to Discontinuation of Study Therapy | 30 |
| 7.6.4 | Adverse Events Leading to Dose Modification | 31 |
| 7.6.5 | Adverse Events | 31 |
| 7.6.6 | Select Adverse Events | 31 |
| 7.6.7 | Immune modulating medication | 31 |
| 7.6.8 | Multiple Events | 31 |
| 7.6.9 | Clinical laboratory evaluations | 31 |
| 7.6.10 | Vital Signs and Pulse Oximetry | 31 |
| 7.6.11 | Immunogenicity Analysis | 31 |
| 7.6.12 | Pregnancy | 31 |
| 7.6.13 | Clinical Safety Program (CSP) | |
| 7.6.14 | Adverse Events by Subgroup | 31 |
| 7.6.15 | Immune-mediated Adverse Events Analysis | 31 |
| 7.7 | Pharmacokinetics | 32 |
| 7.8 | Biomarker Analyses | 32 |
| 7.8.1 | PD-L1 Expression | 32 |
| 7.8.1.1 | Descriptive Statistics of PD-L1 Expression and PD-L1 Status | 32 |

| 7.8.1.2 | Evalua | tion of Associations between PD-L1 Status and Efficacy Measures | 32 |
|---|---|---|---|
| 7.8.1.3 | 1.3 Association of select AE and PD-L1 expression | | |
| 7.9 | Outcon | ne Research Analyses | 33 |
| 7.9.1 | EORTC | EORTC-QLQ-C30 Questionnaire | |
| 7.9.2 | EQ-5D | EQ-5D Questionnaire | |
| 7.10 | Interim | Analysis | 34 |
| 8 | CONV | ENTIONS | 34 |
| 9 | CONTI | ENT OF REPORTS | 35 |
| 10 | DOCU | MENT HISTORY | 35 |
| 11 | REFER | ENCES | 36 |
| Table 2.1 | -1: | Schedule of Spiral CT/MRI Tumor Assessments | |
| Table 2.1 | 1. | LIST OF TABLES Schodula of Spiral CT/MRI Tumor Accessments | 0 |
| Table 2.4 | -1: | Protocol Amendments | |
| Table 4.1 | -1: | 2007 IWG Response Criteria for Malignant Lymphoma | |
| Table 4.2 | .4-1: | Censoring scheme used in primary analysis of PFS | |
| Table 4.3 | .7.1-1: | Time Windows for EORTC-QLQ-C30 Assessments | |
| Table 5-1 | : | Observed ORR with Exact 95% CI | 19 |
| Table 7.4 | .1-1: | Administration of study therapy: definition of parameters | 24 |
| Table 10- | ·1: | Document History | 35 |
| | | LIST OF FIGURES | |
| Figure 2. | 1-1: | Study Design Schematic | 8 |



#### **Research Hypothesis:**

Treatment with nivolumab will lead to clinical benefit, as demonstrated by an improved clinically meaningful objective response rate, including durable responses with substantial magnitude of tumor reduction in subjects with refractory FL who have failed therapy with both rituximab and an alkylating agent.

#### **Schedule of Analyses:**

The final analysis of the primary endpoint will occur at least 12 months after the last enrolled subject's first dose of study therapy. It is anticipated that accrual will last 18 months, with approximately 115 subjects enrolled (90 subjects treated). It is anticipated that the analysis of the primary endpoint will take place approximately 30 months from FPFT. Additional survival analysis will be conducted for up to 5 years beyond analysis of the primary endpoint.

#### 2 STUDY DESCRIPTION

## 2.1 Study Design

This is a single-arm Phase 2 study in subjects ≥ 18 years old with relapsed FL after failure of at least two prior lines of therapy (each containing rituximab and/or an alkylating agent). Approximately 90 subjects will be treated with nivolumab 3mg/kg IV every 2 weeks.

Subjects will undergo screening evaluations to determine eligibility within 28 days prior to first dose. Each 14-day dosing period will constitute a cycle. Radiographic study evaluations will take place in accordance with Table 2.1-1. A PET scan is required at baseline for all subjects, and to confirm a complete response (CR). Baseline assessments should be performed within 28 days prior to the first dose, utilizing spiral CT or MRI. An independent radiology review committee (IRRC) will also be utilized. The primary endpoint of this study is IRRC-assessed objective response rate (ORR), using revised 2007 International Working Group (IWG) Criteria for Malignant Lymphoma criteria. Secondary endpoints include IRRC-assessed duration of response (DOR), as well as complete remission rate (CRR) and PFS as determined by IRRC assessment and ORR based on investigator assessment.

The study design schematic is presented in Figure 2.1-1

Figure 2.1-1: Study Design Schematic



| <b>Table 2.1-1:</b> | Schedule of Spiral CT/MRI Tumor Assessments | | |
|---|---|---|---|
| Time On Study | Assessment<br>Frequency | Assessment Week (day 1 of week shown) | Assessment Window |
| Dose 1 to 8<br>Months | Every 8 weeks | 9, 17, 25, 33 | ± 1 week |
| Month 9 to 2<br>Years | Every 12 weeks | 45, 57, 69, 81, 93 | ± 2 weeks |
| > 2 Years | Every 6 months | 119, 145, 171+ | ±3 weeks |

Note: Once subjects discontinue study therapy by proceeding to allogeneic SCT or ASCT, they will not undergo radiographic assessments as per the frequency described here, but will be followed using the following schedule. Tumor assessment (CR or non-CR) will be assessed by the investigator according to the 2007 IWG criteria and will be required on Day 100, at 6 months, 1 year and every year thereafter from the date of stem cell infusion until the first non-CR after SCT is documented.

## 2.2 Treatment Assignment

After the subject's initial eligibility is established and informed consent has been obtained, the subject must be enrolled into the study by calling an interactive voice response system (IVRS) to obtain the subject number. Every subject that signs the informed consent form must be assigned a subject number in IVRS. Since this is a single arm study, all enrolled subjects who meet eligibility criteria will be treated with nivolumab at 3mg/kg IV every 2 weeks.

## 2.3 Blinding and Unblinding

Not applicable

#### 2.4 Protocol Amendments

This SAP incorporates the following protocol amendments.

**Table 2.4-1:** Protocol Amendments

| Amendments | Date of Issue | <b>Summary of Major Changes</b> |
|---|---|---|
| Revised Protocol Number: 03<br>Incorporates amendment 04 | 21-JUL-2016 | Update of Annex 1 of Protocol Algorithm for safety<br>Management |
| Revised Protocol Number: 02<br>Incorporates amendment 03 | 23-JUL-2014 | Removes the interim analyses and extends the duration of follow-up required for all subjects prior to performing the final analysis of the primary endpoint. |
| | | Modifies a few eligibility criteria to facilitate enrollment. |

**Table 2.4-1:** Protocol Amendments

| Amendments | Date of Issue | Summary of Major Changes |
|---|---|---|
| | | Allows for continued treatment of subjects in certain instances where protocol-defined progression criteria have been met. |
| | | The amendment also serves to clarify various protocol requirements to ensure consistency in the execution of the study including secondary and exploratory objectives, |
| Revised Protocol Number: 01 | 06-Dec-2013 | Per FDA mandatory recommendation: |
| Incorporates amendment(s) 02 and administrative letter 01 | | Exclusion criteria have been added to exclude the following subjects |
| | | Subjects that have received chest radiation ≤ 24 weeks prior to first dose of the study drug |
| | | Additional updates were also made to the protocol including items such as correcting typographical and formatting errors, including errors in the biomarker sampling schedule in Table 5.6-1 |
| Original Protocol | 04-Oct-2013 | Not applicable |

## 2.5 Data Monitoring and Other External Committees

An IRRC will be utilized in this study for determination of IRRC-assessed primary (ORR) and secondary (DOR, CRR, PFS) endpoints. The IRRC will review all available tumor assessment scans for all treated subjects. Details of IRRC responsibilities and procedures will be specified in the IRRC charter.

There will be no data monitoring committee for this study.

#### 3 OBJECTIVES

#### 3.1 Primary objective

To assess the clinical benefit of nivolumab, as measured by independent radiologic review committee (IRRC) assessed objective response rate (ORR) in subjects with FL who have failed therapy with both rituximab and an alkylating agent.

## 3.2 Secondary objectives

- To assess the duration of response (DOR) based on IRRC assessments
- To assess the complete remission rate (CRR) and the duration of CR based on IRRC assessment

- To assess the partial remission (PR) rate and the duration of PR based on IRRC assessment
- To assess progression free survival (PFS) based on IRRC assessment
- To assess the objective response rate (ORR), based on investigator assessments

## 3.3 Exploratory Objectives



#### 4 ENDPOINTS

# 4.1 Primary endpoint ORR (IRRC-assessed)

The primary objective will be measured by the primary endpoint of IRRC-assessed ORR. It is defined as the number of subjects with a best overall response (BOR) of CR or PR, according to the 2007 IWG criteria (see Table 4.1-1), divided by the number of treated subjects. The final analysis of the primary endpoint will occur at least 12 months after the last enrolled subject's first dose of study therapy. The BOR is defined as the best response designation recorded between the date of first dose and the date of initial objectively documented progression per the 2007 IWG criteria or the first subsequent therapy date per IRRC, whichever occurs first.

The first subsequent therapy date per IRRC is determined by the IRRC based on non-palliative radiotherapy, local tumor treatment, systemic anti-cancer therapy and Stem Cell Transplant with a start date on or after the first study therapy date.

For subjects without documented progression or subsequent therapy, all available response designations will contribute to the BOR determination. For purposes of analysis, if a subject receives one dose and discontinues the study without assessment or receives subsequent therapy prior to assessment, this subject will be counted in the denominator (as non-responder).

The IRRC-assessed objective response will be further characterized by the time to response (TTR). TTR is defined as the time from first dosing date to the date of the first response (PR or CR), as assessed by the IRRC.

Table 4.1-1: 2007 IWG Response Criteria for Malignant Lymphoma

| Response | Definition | Nodal masses | Spleen, Liver | Bone marrow |
|---|---|---|---|---|
| CR | Disappearance<br>of all evidence<br>of disease | (a) FDG-avid or PET positive prior to therapy; residual mass of any size permitted if PET negative (b) Variably FDG-avid or PET negative; regression to normal size on CT | Not palpable,<br>nodules<br>disappeared | Infiltrate cleared on<br>repeat biopsy; if<br>indeterminate by<br>morphology,<br>immunohistochemistry<br>should be negative |
| PR | Regression of<br>measurable<br>disease and no<br>new sites | ≥ 50% decrease in SPD of up to 6 largest dominant masses (index lesions); no increase in size of other nodes (non-index lesions) (a) FDG-avid or PET positive prior to therapy; one or more PET positive at previously involved site (b) Variably FDG-avid or PET negative; regression on CT | ≥ 50% decrease<br>in SPD of<br>nodules (for<br>single nodule in<br>greatest<br>transverse<br>diameter); no<br>increase in size<br>of liver or<br>spleen | Irrelevant if positive<br>prior to therapy; cell<br>type should be<br>specified |
| SD | Failure to attain<br>CR/PR or PD | <ul> <li>(a) FDG-avid or PET positive prior to therapy; PET positive at prior sites of disease and no new sites on CT or PET</li> <li>(b) Variably FDG-avid or PET negative; no change in size of previous lesions on CT</li> </ul> | N/A | N/A |
| Relapsed<br>disease<br>or PD | Any new lesion<br>or increase by<br>≥ 50% of<br>previously<br>involved sites<br>from nadir | Appearance of a new lesion(s) > 1.5 cm in any axis, ≥ 50% increase in SPD of more than one node (index lesions), or ≥ 50% increase in longest diameter of a previously identified node > 1cm in short axis. Lesions PET positive if FDG-avid lymphoma or PET positive prior to therapy | > 50% increase<br>from nadir in<br>the SPD of any<br>previous lesions | New or recurrent involvement |

Key: CR = complete remission CT = computed tomography; FDG = [18F] fluorodeoxyglucose; IWG = International Working Group; NA = Not applicable; PD = progressive disease; PET = positron-emission tomography; PR = partial remission; SD = stable disease; SPD = sum of the product of the diameters

## 4.2 Secondary Endpoints

## 4.2.1 Duration of Response (IRRC-assessed)

Duration of response (DOR) is defined as the time from first response (CR or PR) to the date of initial objectively documented progression as determined using the 2007 revised International

Working Group Criteria for Malignant Lymphoma or death due to any cause, whichever occurs first. For subjects who neither progress nor die, the DOR will be censored on the date of their last evaluable tumor assessment. Subjects who start subsequent therapy without a prior reported progression will be censored at the last evaluable tumor assessments prior to or on the first subsequent therapy date per IRRC. This endpoint will only be evaluated in subjects with objective response of CR or PR. Ongoing responders are defined as responders who did not progress, did not die, are not off study and did not started a subsequent therapy.

Duration of Stable Disease will also be evaluated for subjects with SD as best response. Duration of SD is defined as the time between the first dose date to the date of the first documented progression, as determined by IRRC, or death due to any cause, whichever occurs first. Subjects who neither progress nor die will be censored at the same time they will be censored for the DOR analysis.

## 4.2.2 Complete Remission Rate and Duration (IRRC-assessed)

The complete remission rate (CRR) is defined as the number of subjects with a BOR of CR according to the 2007 revised International Working Group Criteria for Malignant Lymphoma, based on IRRC assessment, divided by the number of treated subjects.

To further characterize CRR, the duration of CR will also be evaluated in subjects with objective response of CR. Duration of CR is defined as the time from first documentation of CR (the date of first negative FDG-PET scan or the date of first documentation of no disease involvement in the bone marrow (if required), whichever occurs later) to the date of initial objectively documented progression as determined using the 2007 IWG criteria or death due to any cause, whichever occurs first. Censoring will be applied as per DOR definition.

## 4.2.3 Partial Remission Rate and Duration (IRRC-assessed)

The partial remission rate (PRR) is defined as the number of subjects with a BOR of PR according to the 2007 revised International Working Group Criteria for Malignant Lymphoma, based on IRRC assessment, divided by the number of treated subjects.

To further characterize PRR, the duration of PR will also be evaluated in subjects with objective response of PR. Duration of PR is defined as the time from first documentation of PR to the date of initial objectively documented progression as determined using the 2007 IWG criteria or death due to any cause, whichever occurs first. Censoring will be applied as per DOR definition.

## 4.2.4 Progression Free Survival (IRRC-assessed)

Progression free survival (PFS) is defined as the time from first dosing date to the date of the first documented progression, as determined by an IRRC according to the 2007 revised International Working Group Criteria for Malignant Lymphoma, or death due to any cause, whichever occurs first.

• Subjects who have no baseline tumor assessment will be censored at their first dosing date.

- Subjects who have baseline tumor assessment and who die without a reported progression will be considered to have progressed on the date of their death.
- Subjects who did not progress or die will be considered as not progressed and will be censored on the date of their last assessment.
- Subjects who did not have any on study assessments and did not die will be censored on the first dosing date.
- Subjects who started any subsequent anti-cancer therapy without a prior reported progression will be censored at the last assessment prior to or on their first subsequent therapy date.

Table 4.2.4-1: Censoring scheme used in primary analysis of PFS

| Situation | Date of Progression or Censoring | Outcome |
|---|---|---|
| No baseline tumor assessments | First Dosing date | Not<br>Progressed |
| No on study tumor assessments and no death | First Dosing date | Not<br>Progressed |
| No progression per 2007 IWG criteria and no new anti-cancer treatment started | Date of last tumor assessment with no documented progression per the 2007 IWG criteria | Not<br>Progressed |
| New anticancer treatment started without a prior reported progression per 2007 IWG criteria | Date of last tumor assessment prior or on the date of initiation of the subsequent anti-cancer therapy | Not<br>Progressed |
| Progression per 2007 IWG criteria<br>documented between scheduled visits or at<br>scheduled visit without prior new anticancer<br>treatment started | Date of the first documented tumor progression per<br>the 2007 IWG criteria | Progressed |
| Death without progression per 2007 IWG criteria and without prior new anticancer treatment started | Date of death | Progressed |

To further characterize PFS, progression by response to most recent prior systemic cancer therapy and progression by number of prior systemic cancer therapy lines may also be evaluated.

## 4.2.5 Objective Response Rate (Investigator-assessed)

Investigator-assessed ORR is defined similarly as described for the primary endpoint above (Section 4.1) and will be further characterized by TTR and DOR.

First subsequent therapy date per Investigator is defined as the earliest start date on or after the first study therapy date among systemic anti-cancer therapy, stem cell transplant, non-palliative radiotherapy and local tumor treatment (non-palliative radiotherapy or other).





#### 4.3.7 Outcome Research

#### 4.3.7.1 EORTC-QLQ-C30

Health-related quality of life (HRQoL) will be assessed using the European Organization for Research and Treatment of Cancer (EORTC) QLQ-C30 questionnaire Version 3. It is a 30-item instrument that has gained wide acceptance in oncology clinical studies. The EORTC QLQ-C30 is composed of multi-item and single scales. These include five functional scales (physical, role, emotional, social, and cognitive), three symptom (fatigue, nausea and vomiting, and pain) and a global health status/QOL scale and six single items (dyspnea, insomnia, appetite loss, constipation, diarrhea and financial difficulties). All scales and single items meet the standards for reliability. The reliability and validity of the questionnaire is highly consistent across different language-cultural groups<sup>30</sup>. Except for the overall health status and global quality of life items, responses for all items are 4 point categorical scales ranging from 1 (Not at all) to 4 (Very much). The overall health status/quality of life responses are 7-point Likert scales.

Data will be scored according to the algorithm described in the EORTC QLQ-C30 scoring manual, as follows:

#### **Functional scales:**

- Physical functioning: (1 ((Q1+Q2+Q3+Q4+Q5)/5 1)/3) \* 100
- Role functioning: (1 ((Q6+Q7)/2-1)/3) \* 100
- Emotional functioning: (1 ((Q21+Q22+Q23+Q24)/4-1)/3) \* 100
- Cognitive functioning: (1 ((Q20+Q25)/2-1)/3) \* 100
- Social functioning: (1 ((Q26+Q27)/2-1)/3) \* 100

#### Global health status:

• Global health status/QoL: ((Q29+Q30)/2-1)/6 \* 100

#### **Symptom scales/items:**

- Fatigue: ((Q10+Q12+Q18)/3-1)/3 \* 100
- Nausea and vomiting: ((Q14+Q15)/2-1)/3 \* 100
- Pain: ((O9+O19)/2-1)/3 \* 100

Dyspnea: ((Q8-1)/3 \* 100
Insomnia: (Q11-1)/3 \* 100
Appetite loss: (Q13-1)/3 \* 100
Constipation: (Q16-1)/3 \* 100
Diarrhea: (Q17-1)/3 \* 100

• Financial difficulties: (Q28-1)/3 \* 100

Missing values will be imputed for missing items by "assuming that the missing items have values equal to the average of those items which are present" for any scale in which at least half the items are completed. A scale in which less than half of the items are completed will be treated as missing. This is the method proposed in the scoring manual. A questionnaire will be considered as received if at least one of the 15 scales is non-missing (after imputation).

All questionnaires completed at baseline and on-study will be assigned to a time-point according to the windowing criteria in Table 4.3.7.1-1 and included in the analysis. In case a subject has two on-study assessments within the same window, the assessment closest to the time-point will be used. And, in the case of two assessments at a similar distance to the time-point, the latest one will be chosen. In the event where the subject has no assessment at all in a specific window, the observation will be treated as missing for that time-point.

Table 4.3.7.1-1: Time Windows for EORTC-QLQ-C30 Assessments

| Nominal Time-Point | Time Window |
|-----------------------------|------------------------------------------------|
| Week 1 (Baseline) | Prior to first dose on Day 1 |
| Week 9 | Day 2 thru Day 85, inclusive |
| Every 8 weeks up to week 25 | Nominal Day (+ 28 days / - 27 days, inclusive) |
| Week 33 | Day 198 thru Day 267, inclusive |
| Every 12 weeks thereafter | Nominal Day (+ 42 days / - 41 days, inclusive) |
| Follow-up 1 | NA |
| Follow-up 2 | NA |

#### 4.3.7.2 EuroQoL EQ-5D

Subjects' overall health status will be assessed using the EuroQol Group's self-reported health status measure (EQ-5D-3L)<sup>31</sup>. EQ-5D essentially has 2 components- the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS).

The EQ-5D descriptive system comprises the following 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels: no problems, some problems, severe problems. Once the data have been collected and a database created, a scoring function can be used to assign a value (i.e., EQ-5D index score) to self-reported health states from a set of population-based preference weights.

The EQ VAS records the subject's self-rated health state on a 100-point vertical, visual analogue scale (0 = worst imaginable health state; 100 = best imaginable health state)<sup>32</sup>.



#### 5 SAMPLE SIZE AND POWER

The planned sample size for this study will be approximately 90 treated subjects. The sample size was determined based on two considerations: the ability to produce a CI which would exclude an ORR of 20%, which is not considered clinically relevant and provide sufficient information for a reliable understanding of the safety profile.

Assuming the true ORR is 35%, the study has approximately 87% power to reject the null hypothesis that the true ORR is  $\leq$  20%, considering a 2-sided alpha of 5%. In addition, Table 5-1 summarizes the 95% exact CI for the target ORRs ranging from 30% to 44% with sample size of 90. At observed ORR  $\geq$  30%, the lower bound of the 95% CI excludes 20%.

| 1 able 5-1: | Observed ORR with Exact 95% ( | I۔ |
|-------------|-------------------------------|----|

| True ORR | 95% Exact CI |
|----------|---------------|
| 30% | [20.8%-40.6%] |
| 34% | [24.7%-45.2%] |
| 40% | [29.8%-50.9%] |
| 44% | [34.0%-55.3%] |

# 6 STUDY PERIODS, TREATMENT REGIMENS AND POPULATIONS FOR ANALYSES

# 6.1 Study Periods

#### 6.1.1 Baseline Period

Baseline evaluations or events will be defined as evaluations or events that occur before the date and time of the first dose of study treatment.

In cases where the time (onset time of event or evaluation time and dosing time) is missing or not collected, the following definitions will apply:

- Pre-treatment AEs will be defined as AEs with an onset date prior to but not including the day of the first dose of study treatment
- Baseline evaluations (laboratory tests, pulse oximetry and vital signs) will be defined as evaluations with a date on or prior to the day of first dose of study treatment

If there are multiple valid assessments, the assessment that is closest to day (and time if collected) of the first dose of study treatment will be used as the baseline in the analyses. If multiple

assessments are collected at the same date (and time if collected), the assessment with the latest database entry date (and time if collected) will considered as baseline.

#### 6.1.2 Post Baseline Period

On-treatment AEs will be defined as AEs with an onset date-time on or after the date-time of the first dose of study treatment (or with an onset date on or after the day of first dose of study treatment if time is not collected or is missing). An AE will be counted as on-treatment if the event occurred within 30 days (or 100 days depending on analysis) of the last dose of study treatment. Refer to Core SAP<sup>29</sup>.

On-treatment evaluations (laboratory tests, pulse oximetry and vital signs) will be defined as evaluations taken after the day (and time, if collected and not missing) of first dose of study treatment. An evaluation will be counted as on-treatment if it occurred within 30 days (or 100 days depending on analysis) of the last dose of study treatment. Refer to Core SAP<sup>29</sup>.

## 6.2 Treatment Regimens

All subjects will be treated with nivolumab.

## 6.3 Populations for Analyses

## 6.3.1 Analysis Populations

The following populations will be defined.

- All enrolled subjects: All subjects who signed an informed consent form and were registered into the IVRS.
- All treated subjects: All enrolled subjects who received at least one dose of nivolumab. This is the primary population for efficacy and safety.
- All response evaluable subjects: All treated subjects who have baseline and at least one onstudy evaluable tumor measurement.
- **PK subjects**: All enrolled subjects with available serum time-concentration data from subjects dosed with nivolumab.
- **Immunogenicity evaluable subjects**: all treated subjects with baseline and at least one post baseline immunogenicity assessment.
- All PD-L1 tested subjects: All enrolled subjects who had a tumor tissue sample available for assessment of PD-L1 expression.
- All PD-L1 evaluable subjects: All treated subjects with quantifiable baseline PD-L1 expression
- **Biomarker subjects**: All treated subjects with available biomarker data.
- Outcomes Research subjects: all treated subjects who have an assessment at baseline (Visit 1 assessment prior to administration of drug) and at least 1 subsequent assessment (for EORTC QLQ-C30 and EQ-5D separately).

#### 7 STATISTICAL ANALYSES

#### 7.1 General Methods

Unless otherwise noted, the bulleted titles in the following subsections describe tabulations of discrete variables, by the frequency and proportion of subjects falling into each category. Percentages given in these tables will be rounded and, therefore, may not always sum to 100%. Continuous variables will be summarized using the mean, standard deviation, median, minimum and maximum values.

Time to event distribution (e.g. progression free survival, overall survival, time to response, and duration of response) will be estimated using Kaplan Meier techniques. Median survival time along with 95% CI will be constructed based on a log-log transformed CI for the survivor function  $S(t)^{33,34}$ . Rates at fixed time points will be derived from the Kaplan Meier estimate and corresponding confidence interval will be derived based on Greenwood formula<sup>35</sup> for variance derivation and on log-log transformation applied on the survivor function  $S(t)^{36}$ .

## 7.2 Study Conduct

#### 7.2.1 Accrual

The following will be summarized on the enrolled population:

- Number of subjects accrued by country and investigational site
- Number of subjects accrued by month

A by subject listing of accrual will be produced.

#### 7.2.2 Relevant Protocol Deviations

The following programmable deviations will be considered as relevant protocol deviations. Non-programmable relevant eligibility and on-treatment protocol deviations, as well as significant (both programmable and non-programmable) eligibility and on-treatment protocol deviations will be reported through ClinSIGHT listings.

#### At entrance:

- Subjects without documented relapsed or refractory FL.
- Subjects without treatment of FL consisting of ≥ 2 prior treatment lines; each of the two prior treatment lines must include a CD20 and/or an alkylating agent (e.g., bendamustine, cyclophosphamide, ifosfamide, chlorambucil, melphalan, busulfan, nitrosoureas). At least one of the prior treatment lines must include rituximab.
- Subject without measurable disease at baseline.
- Subject with baseline ECOG not in (0, 1).

#### **On-Study:**

• Any concurrent antineoplastic therapy (i.e., chemotherapy, hormonal therapy, immunotherapy, radiation therapy except for palliative radiation therapy, or standard or investigational agents for treatment of cancer).

A by subject listing will be produced.

## 7.3 Study Population

#### 7.3.1 Subject Disposition

The total number of subjects enrolled (treated or not) will be presented along with the reason for not being treated.

Number of subjects who discontinued treatment along with corresponding reason will also be tabulated.

## 7.3.2 Demographics and Other Baseline Characteristics

Descriptive statistics will be summarized the following baseline characteristics for all treated subjects. All baseline presentations will identify subjects with missing measurements. Listings will also be provided.

- Age (descriptive statistics)
- Age categories ( $< 65, \ge 65 \text{ and } < 75, \ge 75$ )
- Gender, Race/Ethnicity
- Region (US/Canada vs. Europe vs. Rest of World)
- ECOG PS (0, 1, >1, Not Reported)
- weight
- Smoking Status (current/former vs never smoker vs. unknown)
- Time from initial disease diagnosis to first dose of nivolumab (descriptive statistics and  $(< 1 \text{ year}, 1 < 2 \text{ year}, 2 < 3 \text{ year}, 3 < 5 \text{ year}, 5 < 7 \text{ year}, 7 < 10 \text{ year}, \ge 10 \text{ years})$
- Disease stage at initial diagnosis (Stage I-II-III-IV)
- Follicular lymphoma international prognostic index (FLIPI) Score (0, 1, 2, 3, 4, 5) at initial diagnosis
- Lymphoma involvement in bone marrow at baseline (Yes/No/Not Reported)
- Disease status at study entry (Relapse, Refractory)
- All lesions (Investigator Tumor Assessments at Baseline): sites of diseases, number of disease sites per subject
- Target Lesions (Investigator Tumor Assessments at Baseline): Presence of target lesions, site of target lesion, sum of diameters of target lesions.

#### 7.3.3 Medical History

General medical history will be listed by subject and pretreatment events will be tabulated.

## 7.3.4 Prior therapy

The following will be summarized:

- Number of subjects by type of prior therapy received:
  - Immunotherapy by Monoclonal Antibodies
  - Steroid
  - Chemotherapy Anthracyclines
  - Chemotherapy Other than Anthracyclines
  - Kinase Inhibitors
  - Immunomodulary Derivatives
  - Radioimmunotherapy
  - Other
- Number of subjects per type of regimen for first line of therapy (e.g. R-CHOP vs R-CVP vs OTHER)
- Number of prior systemic cancer therapy lines received  $(0, 1, 2, 3, 4, \ge 5)$
- Best response to most recent prior systemic cancer therapy (CR vs. PR vs. SD vs. Relapse/PD vs. Unable to Determine vs. Not Applicable vs. Not Reported) (Note: Not Applicable is used when the agent is a conditioning regimen for stem cell transplant)
- Time from completion of most recent prior regimen to treatment (< 3, 3 6, > 6 months)
- Prior radiotherapy (yes, no)
- Prior autologous transplant (yes, no)

Other Prior therapy:

• Prior/current non-study medication classified by anatomic and therapeutic classes.

Medication will be reported using the generic name. A listing by subject will also be provided.

#### 7.3.5 Baseline Examinations

Percentage of subjects with abnormal baseline physical examination will be tabulated by examination criteria.

## 7.4 Extent of Exposure

Analyses in this section will be performed in all treated subjects.

## 7.4.1 Administration of Study Therapy

The following parameters will be summarized (descriptive statistics):

- Relative dose intensity (%) using the following categories: < 50%; 50 < 70%; 70 < 90%; 90 < 110%; ≥ 110%.</li>
- Number of doses received (summary statistics)
- Cumulative dose
- Duration of treatment: duration of treatment will be presented using a Kaplan-Meier curve whereby the last dose date will be the event date for subjects who discontinued study therapy. Subjects who are still on study therapy will be censored on their last dose date. Median duration of treatment and associated 95% CI will be provided.
- A by-subject listing of dosing of study medication (record of study medication, infusion details, dose change) and a listing of batch number will be also provided.

Table 7.4.1-1: Administration of study therapy: definition of parameters

| | nivolumab |
|---|---|
| Dosing schedule per protocol | 3mg/kg every 2 weeks |
| Dose | Dose (mg/kg) is defined as Total Dose administered (mg)/Most recent weight (kg). Dose administered in mg at each dosing date and weight are collected on the CRF. |
| Cumulative Dose | Cum dose (mg/kg) is sum of the doses (mg/kg) administered to a subject during the treatment period. |
| Relative dose intensity (%) | Cum dose (mg/kg) / [ (Last dose date - Start dose date + 14) x 3 /14 ] x 100 |
| Duration of treatment | Last dose date - Start dose date + 1 |

## 7.4.2 Modifications of Study Therapy

#### 7.4.2.1 Dose delays

Treatment may be delayed for up to a maximum of 6 weeks from the last dose. A dose will be considered as actually delayed if the delay is exceeding 3 days (i.e., greater than or equal to 4 days from scheduled dosing date). Length of delay is defined as (duration of previous cycle in days - 14). Dose delays will be divided into following categories: 4 - < 8 days, 8 - < 15 days, 15 - < 42,  $\ge 42$  days. Reason for dose delay/omission will be retrieved from CRF dosing pages.

The following parameters will be summarized.

• Number of subjects with at least one dose delayed, number of dose delayed per subject, Length of Delay and Reason for Dose Delay

### 7.4.2.2 Infusion Interruptions and Rate Changes

The following parameters will be summarized:

• Number of subjects with at least one dose infusion interruption, number of infusion interruptions per subject and the reason for interruption.

• Number of subjects with at least one IV infusion rate reduction, number of IV infusion rate reduction per subject and the reason for reduction

#### 7.4.2.3 Dose Reductions/Escalation

There will be no dose escalations or reductions of nivolumab allowed.

#### 7.4.3 Concomitant Medications

Concomitant medications, defined as medications other than study medications which are taken at any time on-treatment (i.e. on or after the first day of study therapy and within 100 days following the last dose of study therapy), will be coded using the WHO Drug Dictionary.

The following summary tables will be provided:

• Concomitant medications (subjects with any concomitant medication, subjects by medication class and generic term).

A by-subject listing will accompany the table.

## 7.5 Efficacy

## 7.5.1 Primary endpoint of ORR (IRRC-assessed)

The IRRC-assessed ORR (using revised IWG Criteria for Malignant Lymphoma criteria) will be summarized on the all subjects treated population by a binomial response rate. The Clopper-Pearson<sup>37</sup> method will be used to estimate the two-sided 95% CI.

BOR will be summarized by response category.

Summary statistics of time to objective response will be provided for subjects who achieve PR or CR, as assessed by the IRRC. CR requires confirmation by PET. To assess tumor response kinetics, time to response will also be analyzed using the KM methodology for all treated subjects. Kaplan-Meier curve will represent the cumulative rate of response over time. For the non-responders, time to response will be censored at the maximum time of response + 1 day of all subjects. Cumulative Response Rates will be tabulated for Week 9, Month 4, 6, 8, 12 and 18, and overall Response Rate will be provided.

### 7.5.1.1 ORR Subgroups

To assess consistency of ORR, IRRC-assessed ORR (primary analysis) will be summarized for the following subgroups:

- Age  $(<65, \ge 65 \text{ and } < 75, \ge 75)$
- Region (US/Canada, Europe, Rest of the world).
- Gender (Male, Female)
- Race (White, Black or African American, Asian, and Other (pooling all other possibilities)
- Smoking status (current/former vs never smoker vs unknown)

- ECOG (0, 1, >1, NOT REPORTED)
- Number of prior therapies  $(0, 1, 2, 3, 4, \ge 5)$
- Prior Autologous Transplant (Yes, No)
- Time from most recent prior systemic cancer therapy to first dose of nivolumab (< 3 months, 3 6 months, > 6 months)
- Refractory, Relapsed Lymphoma (which is the disease diagnosis status at study entry)
- FLIPI Score (0-1, 2, 3, 4-5)

Categories including less than 5 subjects may be collapsed. Analyses of subgroups of less than 5 subjects may not be provided.

## 7.5.1.2 Sensitivity analyses for ORR

- As sensitivity analysis, a summary of IRRC-assessed ORR based on response evaluable subjects instead of all treated subjects will also be presented. Clopper Pearson 95% CI will be used in this analysis.
- To assess concordance between IRRC (primary analysis) and investigator assessments, BOR
  will be cross-tabulated by assessment type (Investigator vs IRRC). Concordance Rate of
  Responders will be computed as the frequency with which Investigator and IRRC agree on
  classification of a subject as responder/non responder as a proportion of the total number of
  subjects assessed.

## 7.5.2 Secondary Endpoint of Duration of Response (IRRC-assessed)

The DOR will be summarized for subjects who achieve PR or CR as determined by IRRC using KM product-limit method. Two-sided, 95% confidence intervals for median DOR will be constructed based on log-log transformation. Range of duration of response and the number of ongoing responders will also be presented. In addition, the percentage of responders still in response at different time points (3, 6 and 12 months) will be presented based on the DOR KM plot.

The status of subjects who are censored in the duration of response analysis will be tabulated using the following categories:

- received subsequent anti-cancer therapy
- off-study (with reason)

Duration of stable disease will also be estimated using KM product-limit method for subjects with SD as best response. Two-sided, 95% confidence intervals for median duration of SD will be computed.

# 7.5.3 Secondary Enpoint of Complete Remission Rate (IRRC-assessed)

IRRC-assessed CRR will be summarized by a binomial response rate and its corresponding two-sided 95% exact CIs using the Clopper-Pearson<sup>37</sup> method.

To further characterize CRR, the duration of CR will be summarized for subjects who achieve CR as determined by IRRC using KM product-limit method. Two-sided, 95% confidence intervals for median duration of CR will be constructed based on log-log transformation. Range of duration of CR will also be presented.

# 7.5.4 Secondary Endpoint of Partial Remission Rate and Duration (IRRC-assessed)

IRRC-assessed PRR will be summarized by a binomial response rate and its corresponding two-sided 95% exact CIs using the Clopper-Pearson<sup>31</sup> method.

To further characterize PRR, the duration of PR will be summarized for subjects who achieve PR as determined by IRRC using KM product-limit method. Two-sided, 95% confidence intervals for median duration of PR will be constructed based on log-log transformation. Range of duration of PR will also be presented.

## 7.5.5 Secondary Endpoint of Progression Free Survival (IRRC-assessed)

IRRC-assessed PFS will be summarized descriptively using the Kaplan-Meier (KM) product-limit method. Median values of PFS, along with two-sided 95% CIs (based on the log-log transformation), will also be calculated.

The source of progression (death vs. progression) will be summarized.

The status of subjects who are censored in the PFS Kaplan-Meier analysis will be tabulated using following categories:

- Received subsequent anti-cancer therapy (Stem Cell Transplant, other)
- Still on-treatment
- Progression-free in follow-up
- Off-study: (lost to follow-up, withdrew consent, other).

KM curve of PFS will be generated. PFS rates per IRRC at 6, 9 and 12 months will be estimated using KM estimates on the PFS curve. PFS rates at 18, 24 and 36 months may also be estimated depending on whether minimum follow-up will be longer than timepoint to generate the rate. Associated two-sided 95% CIs will be calculated.

KM curves of PFS by response of most recent prior systemic cancer therapy as well as KM curves of PFS by number of prior systemic anti-cancer therapy lines will also be generated. Some categories may be collapsed to have sufficient number of subjects in each category. Median values of PFS in each category along with two-sided 95% CIs (based on the log-long transformation) will also be calculated.

# 7.5.6 Secondary Endpoint of Objective Response Rate (Investigator-assessed)

Investigator-assessed ORR will be summarized by a binomial response rate and its corresponding two-sided 95% exact CIs using the Clopper-Pearson<sup>37</sup> method<sup>37</sup>

Investigator-assessed BOR will be summarized by response category.

Summary statistics of time to objective response will be provided for subjects who achieve PR or CR, as assessed by the Investigator. CR requires confirmation by PET. To assess tumor response kinetics, time to response will also be analyzed using the KM methodology for all treated subjects. Kaplan-Meier curve will represent the cumulative rate of response over time. For the non-responders, time to response will be censored at the maximum time of response + 1 day of all subjects. Cumulative Response Rates will be tabulated for Week 9, Month 4, 6, 8, 12 and 18, and overall Response Rate will be provided.







# 7.6 Safety

All analyses from the Core Safety SAP<sup>29</sup> will be produced.

# 7.6.1 Deaths

See Core Safety SAP<sup>29</sup>.

# 7.6.2 Serious Adverse Events

See Core Safety SAP<sup>29</sup>.

# 7.6.3 Adverse Events Leading to Discontinuation of Study Therapy

See Core Safety SAP<sup>29</sup>.

## 7.6.4 Adverse Events Leading to Dose Modification

See Core Safety SAP<sup>29</sup>.

#### 7.6.5 Adverse Events

See Core Safety SAP<sup>29</sup>

#### 7.6.6 Select Adverse Events

See Core Safety SAP<sup>29</sup>

## 7.6.7 Immune modulating medication

See Core Safety SAP<sup>29</sup>.

## 7.6.8 Multiple Events

See Core Safety SAP<sup>29</sup>.

## 7.6.9 Clinical laboratory evaluations

See Core Safety SAP<sup>29</sup>.

## 7.6.10 Vital Signs and Pulse Oximetry

See Core Safety SAP<sup>29</sup>.

# 7.6.11 Immunogenicity Analysis

See Core Safety SAP<sup>29</sup>.

# 7.6.12 Pregnancy

By-subject listing of pregnancy tests results will be provided

# 7.6.13 Clinical Safety Program (CSP)

See Core Safety SAP<sup>29</sup>.

## 7.6.14 Adverse Events by Subgroup

See Core Safety SAP<sup>29</sup>.

# 7.6.15 Immune-mediated Adverse Events Analysis

See Core Safety SAP<sup>29</sup>.

#### 7.7 Pharmacokinetics

The nivolumab concentration data obtained in this study may be combined with data from other studies in the clinical development program to develop or refine a population PK model. This model may be used to evaluate the effects of intrinsic and extrinsic covariates on the PK of nivolumab and to determine measures of individual exposure (such as steady-state peak, trough, and time-averaged concentration). In addition, model determined exposures may be used for exposure-response analyses. Results of population PK and exposure response-analyses will be reported separately.





## 7.9 Outcome Research Analyses

#### 7.9.1 EORTC-QLQ-C30 Questionnaire

Unless otherwise specified, the analysis of EORTC QLQ C-30 will be performed in all treated subjects who have an assessment at baseline and at least one subsequent assessment. Analyses will be performed.

Baseline measures will be summarized using descriptive statistics (N, mean, standard deviation, median, first and third quartiles, minimum, maximum) for each QLQ-C30 item, as well as global and functional scales, based on subjects with a baseline measurement.

Change from baseline will be summarized using descriptive statistics (N, mean, standard deviation, median, first and third quartiles, minimum, maximum) for each QLQ-C30 item, as well as global and functional scales at each assessment time point. In addition, the percentage of subjects demonstrating a clinically meaningful deterioration (defined as a 10 point change from baseline) will be presented for each scale at each assessment timepoint. Percentages will be based on number subjects assessed at baseline and at assessment time point.

EORTC-QLQ-C30 questionnaire completion rate, defined as the proportion of questionnaires actually received out of the expected number (i.e., number of subjects on treatment or in follow up), will be calculated and summarized for each assessment time point.

A by subject listing of QLQ-C30 with each QLQ-C30 item, functional scales and global health status will be provided.

#### 7.9.2 EQ-5D Questionnaire

Unless otherwise specified, the analysis of EQ-5D will be performed in all treated subjects who have an assessment at baseline and at least one subsequent assessment. Analyses will be performed.

Subject's overall health state on a visual analog scale (EQ-VAS) at each assessment time point will be summarized using descriptive statistics (N, mean, SD, median, 25<sup>th</sup> and 75<sup>th</sup> percentiles, minimum, maximum).

Proportion of subjects reporting problems for the 5 EQ-5D dimensions at each assessment time point will be summarized by level of problem. Percentages will be based on number subjects assessed at assessment time point.

A by-subject listing of EQ-5D with the problem levels for each of the 5 dimensions (mobility, self-care, usual activities, pain/discomfort and anxiety/depression), health state (5 dimensions digits combined in a 5-digit number) and EQ-VAS will be provided.

Results of EQ5D-Index will be presented separately and will be described in the GHEOR SAP.

#### 7.10 Interim Analysis

No interim analysis planned. Interim analyses may be conducted if it is necessary in order to make decisions regarding further development. Summaries and listings of efficacy and safety will be provided. Interim analyses will not impact the study duration and the trial will continue as planned.

#### 8 CONVENTIONS

The following conventions may be used for imputing partial dates for analyses requiring dates:

For missing and partial adverse event onset dates, imputation will be performed using the Adverse Event Domain Requirements Specification<sup>38</sup>. Missing and partial Non-Study Medication Domain dates will be imputed using the derivation algorithm described in BMS Non-Study Medication Domain Requirements Specification<sup>39</sup>.

## For death dates, the following conventions will be used for imputing partial dates:

- If only the day of the month is missing, the 1<sup>st</sup> of the month will be used to replace the missing day. The imputed date will be compared to the last known alive date and the maximum will be considered as the death date.
- If the month or the year is missing, the death date will be imputed as the last known alive date
- If the date is completely missing but the reason for death is present the death date will be imputed as the last known alive date

# For date of progression, the following conventions will be used for imputing partial dates:

- If only the day of the month is missing, the 1<sup>st</sup> of the month will be used to replace the missing day.
- If the day and month are missing or a date is completely missing, it will be considered as missing.

• In case, the date of death is present and complete, the imputed progression date will be compared to the date of death. The minimum of the imputed progression date and date of death will be considered as the date of progression.

#### For other partial/missing dates, the following conventions will be used:

- If only the day of the month is missing, the 15th of the month will be used to replace the missing day.
- If both the day and the month are missing, "July 1" will be used to replace the missing information.
- If a date is completely missing, it will be considered as missing.

The following conversion factors will be used to convert days to months or years: 1 month = 30.4375 days and 1 year = 365.25 days.

Duration (e.g. time from first diagnosis to first dosing date, duration response, and time to response) will be calculated as follows:

Duration = (Last date - first date + 1)

All statistical analyses will be carried out using SAS (Statistical Analysis System software, SAS Institute, North Carolina, USA) unless otherwise noted.

#### 9 CONTENT OF REPORTS

All analyses described in the SAP will be included in the Clinical Study Report(s) except where otherwise noted. Refer to the Data Presentation Plan for mock-ups of all tables, figures and listings

#### 10 DOCUMENT HISTORY

Table 10-1: Document History

| Version Number | Author(s) | Description |
|---|---|---|
| 1.0 | Cécile Dorange | Initial version 13-May-2014 |
| 2.0 | Anne Sumbul | Updated on 25-Sep-2015 |
| 3.0 | Anne Sumbul | Updated on 24-Apr-2017 Reference to Protocol v3 (21JUL16) Clarify PFS censoring scheme Addition of definition of ongoing responder Add PFS and OS rate at 9 and 36 months |
| | | <ul> <li>Add Time to Next Treatment</li> <li>Add PFS by response to most recent prior systemic cancer therapy</li> </ul> |

**Table 10-1: Document History** Add PFS by number of prior systemic cancer therapy line Clarify management of raw PD-L1 result = "<1%" Analysis of IMAE is now referring to nivo core safety SAP Clarify notion of subsequent therapy Updated on 27-Jun-2017 3.1 Anne Sumbul Removed "not reported" for prior transplant and prior radiotherapy Add "Not Applicable" to the codelist of best response to prior systemic cancer therapy Add R-CVP as category for first line therapy

#### 11 REFERENCES

- Howlader N, Noone AM, Krapcho M, Garshell J, Neyman N, Altekruse SF, Kosary CL, Yu M, Ruhl J, Tatalovich Z, Cho H, Mariotto A, Lewis DR, Chen HS, Feuer EJ, Cronin KA (eds). SEER Cancer Statistics Review, 1975-2010, National Cancer Institute. Bethesda, MD, http://seer.cancer.gov/csr/1975\_2010/, based on November 2012 SEER data submission, posted to the SEER web site, 2013.
- Armitage JO, Weisenburger DD. New approach to classifying non-Hodgkin's lymphomas: Clinical features of the major histologic subtypes: Non-Hodgkin's Lymphoma Classification Project. J Clin Oncol 1998;16:2780-2795.
- Horning SJ, Rosenberg SA. The natural history of initially untreated low-grade non-Hodgkin's lymphomas. N Engl J Med 1984;311:1471-1475.

- Horning SJ. Natural history of and therapy for the indolent non-Hodgkin's lymphomas. Semin Oncol 1993;20:75-88.
- Villa D, Crump M, Panzarella T, et al. Autologous and allogeneic stem-cell transplantation for transformed follicular lymphoma: a report of the Canadian blood and marrow transplant group. J Clin Oncol. 2013;31(9):1164-71.
- Ardeshna KM, Smith P, Norton A. Long-term effect of a watch and wait policy versus immediate systemic treatment for asymptomatic advanced-stage non-Hodgkin lymphoma: A randomised controlled trial. Lancet 2003;362:516-522.
- Al-Tourah AJ, Gill KK, Chhanabhai M, et al. Population-based analysis of incidence and outcome of transformed non-Hodgkin's lymphoma. J Clin Oncol 2008;26:5165-5169.
- Montoto S, Davies AJ, Matthews J, et al. Risk and clinical implications of transformation of follicular lymphoma to diffuse large B-cell lymphoma. J Clin Oncol 2007;25:2426-2433.
- Mac Manus MP and Hoppe RT. Is radiotherapy curative for stage I and II low-grade follicular lymphoma? Results of a long-term follow-up study of patients treated at Stanford University. J Clin Oncol 1996;14(4):1282–1290.
- Wilder RB, Jones D, Tucker SL, et al. Long-term results with radiotherapy for stage I-II follicular lymphomas. Int J Radiat Oncol Biol Phys 2001;51:1219–1227.
- Brice P, Bastion Y, Lepage E, et al. Comparison in low-tumor-burden follicular lymphomas between an initial no-treatment policy, prednimustine, or interferon alfa: A randomized study from the Groupe d'Etude des Lymphomes Folliculaires: Groupe d'Etude des Lymphomes de l'Adulte. J Clin Oncol 1997;15:1110-1117.
- Gallagher CJ, Gregory WM, Jones AE, et al. Follicular lymphoma: Prognostic factors for response and survival. J Clin Oncol 1986;4:1470-1480.
- McLaughlin P, Grillo-Lopez AJ, Link BK, et al. Rituximab chimeric anti-CD20 monoclonal antibody therapy for relapsed indolent lymphoma: Half of patients respond to a four-dose treatment program. J Clin Oncol 1998;16:2825-2833.
- Czuczman MS, Grillo-Lopez AJ, White CA, et al. Treatment of patients with low-grade B-cell lymphoma with the combination of chimeric anti-CD20 monoclonal antibody and CHOP chemotherapy. J Clin Oncol 1999;17:268-276.
- Marcus R, Imrie K, Belch A, et al. CVP chemotherapy plus rituximab compared with CVP as first-line treatment for advanced follicular lymphoma. Blood 2005;105:1417-1423.
- Herold M, Haas A, Srock S, et al. Rituximab added to first-line mitoxantrone, chlorambucil, and prednisolone chemotherapy followed by interferon maintenance prolongs survival in patients with advanced follicular lymphoma: An East German Study Group Hematology and Oncology Study. J Clin Oncol 2007;25:1986–1992.
- Hiddemann W, Kneba M, Dreyling M, et al. Frontline therapy with rituximab added to the combination of cyclophosphamide, doxorubicin, vincristine, and prednisone (CHOP) significantly improves the outcome for patients with advanced-stage follicular lymphoma

- compared with therapy with CHOP alone: Results of a prospective randomized study of the German Low-Grade Lymphoma Study Group. Blood 2005;106:3725–3732.
- Rummel MJ, Niederle N, Maschmeyer G, et al. On behalf of the Study group indolent Lymphomas (StiL). Bendamustine plus rituximab versus CHOP plus rituximab as first-line treatment for patients with indolent and mantle-cell lymphomas: an open-label, multicentre, randomised, phase 3 non-inferiority trial. The Lancet 2013;381(9873):1203-1210.
- van Oers MH, Klasa R, Marcus RE, et al. Rituximab maintenance improves clinical outcome of relapsed/resistant follicular non-Hodgkin lymphoma in patients both with and without rituximab during induction: Results of a prospective randomized phase 3 intergroup trial. Blood 2006;108:3295-3301.
- <sup>20</sup> Tan D, Horning SJ, Hoppe RT, et al. Improvements in observed and relative survival in follicular grade 1-2 lymphoma during 4 decades: the Stanford University experience. Blood. 2013;Aug 8;122(6):981-7.
- <sup>21</sup> Schnell R, Barth S, Diehl V, Engert A. Non-Hodgkin's Lymphoma: A Review of Immunotherapeutic Approaches to Treatment. BioDrugs 1997;8(3):216-34.
- Kasamon YL, Ambinder RF. Immunotherapies for Hodgkin's lymphoma. Crit Rev Oncol Hematol. 2008;66(2):135-44.
- <sup>23</sup> Cheson, BD and Leonard JP. Monoclonal Antibody Therapy for B-Cell Non-Hodgkin's Lymphoma. N Engl J Med 2008;359:613-626.
- Younes A, Bartlett NL, Leonard JP, et al. Brentuximab Vedotin (SGN-35) for Relapsed CD30-Positive Lymphomas. N Engl J Med 2010;363:1812-1821.
- Mellman I, Coukos G, Dranoff G. Cancer immunotherapy comes of age. Nature 2011; Dec 22;480:480-89.
- <sup>26</sup> Chen DS, Mellman I. Oncology meets immunology: the cancer-immunity cycle. Immunity. 2013;39(1):1-10.
- <sup>27</sup> Brahmer JR, Drake CG, Wollner I, et al. Phase I Study of Single-Agent Anti-Programmed Death-1 (MDX-1106) in Refractory Solid Tumors: Safety, Clinical Activity, Pharmacodynamics, and Immunologic Correlates. J Clin Oncol. 2010;28:3167-3175.
- Topalian SL, Hodi FS, Brahmer JR, et al. Safety, Activity, and Immune Correlates of Anti-PD-1 Antibody in Cancer. The New England Journal of Medicine 2012;366:2443-2454.
- <sup>29</sup> Core Safety Statistical Analysis Plan for CA209, Bristol-Myers Squibb.
- Aaronson N.K., Ahmedzai S., et al. The European Organisation for Research and Treatment of Cancer QLQ-30: a quality-of-life instrument for use in international clinical trials in oncology. J Natl Cancer Inst, 85: 365-376, 1993.
- http://www.euroqol.org/about-eq-5d/publications/user-guide.html.
- The EuroQol Group: EuroQol: A new facility for the measurement of health-related quality of life—The EuroQol Group. Health Policy 16:199-208, 1990.

- Brookmeyer R. and Crowley J. A confidence interval for the median survival time. Biometrics 38:29-41, 1982.
- Klein, J. P. and Moeschberger, M. L. (1997), Survival Analysis: Techniques for Censored and Truncated Data, New York: Springer-Verlag.
- Greenwood, M. The errors of sampling of the survivorship tables, Reports on Public Health and Statistical Subjects, 33, Appendix 1, HMSO, London, 1926.
- Kalbfleisch, J. D. and Prentice, R. L. (1980), The Statistical Analysis of Failure Time Data, New York: John Wiley & Sons.
- <sup>37</sup> Clopper, CJ and Pearson, ES. The use of confidence or fiducial limits illustrated in the case of the binomial. Biometrika 26: 404-413, 1934
- Adverse Event Domain Requirements Specification. Bristol-Myers Squibb Co. PRI. Version 2.1.2, April 23, 2012.
- Non-Study Medication Domain Requirements Specification. Bristol-Myers Squibb, Co. PRI. Version 2.2 April 24, 2012.